CLINICAL TRIAL: NCT04271956
Title: A Prospective, Open-label, Multicenter Phase-II Trial to Evaluate the Efficacy and Safety of Zanubrutinib (BGB-3111), a BTK Inhibitor, Plus Tislelizumab (BGB-A317), a PD1 Inhibitor, for Treatment of Patients with Richter Transformation with or Without Sonrotoclax（BGB-11417), a Bcl-2 Inhibitor (CLL-RT1-trial of the GCLLSG).
Brief Title: Efficacy and Safety of Zanubrutinib Plus Tislelizumab Treatment with or Without Sonrotoclax for Patients with Richter Transformation
Acronym: CLL-RT1
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: German CLL Study Group (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLL-RT1; 2023-504653-12-00 (EU CTIS Number)
Record Dates: First submitted 2020-02-14; First posted 2020-02-17 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Richter Transformation
MeSH Terms: interventions — tislelizumab; zanubrutinib

STUDY DESIGN:
Intervention Model Description: Recruitment in cohort 1 (double combination therapy) has already been completed. Recruitment in new cohort 2 (triple combination therapy) will start in Q3 2024.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tislelizumab + Zanubrutinib (Experimental): Induction: 6 cycles (q21d) of Tislelizumab + Zanubrutinib
  Consolidation: 6 cycles (q21d) of Tislelizumab + Zanubrutinib
  Maintenance: Patients with response to therapy continue to take Tislelizumab + Zanubrutinib (Q3W) until disease progression, non-tolerance or when receiving allogeneic stem cell transplantation (SCT) for consolidation
  Interventions: Biological: Tislelizumab; Drug: Zanubrutinib
- Tislelizumab + Zanubrutinib + Sonrotoclax (Experimental): Induction: 6 cycles (q21d) of Tislelizumab + Zanubrutinib + Sonrotoclax
  Consolidation: 6 cycles (q21d) of Tislelizumab + Zanubrutinib + Sonrotoclax
  Maintenance: Patients with response to therapy continue to take Tislelizumab + Zanubrutinib (Q3W) + Sonrotoclax until disease progression, non-tolerance or when receiving allogeneic stem cell transplantation (SCT) for consolidation
  Interventions: Biological: Tislelizumab; Drug: Zanubrutinib; Drug: Sonrotoclax

INTERVENTIONS:
Biological: Tislelizumab — Cycle (q21d): Day 1: Tislelizumab i.v. 200 mg
  Other Names: BGB-A317
Drug: Zanubrutinib — Cycle (q21d): Zanubrutinib p.o. 160 mg twice a day
  Other Names: BGB-3111
Drug: Sonrotoclax — Cycle 1: Sonrotoclax Start Ramp-up to 320 mg QD po Days 1-2 Sonrotoclax 2 mg (2 tabl. at 1mg) Days 3-4 Sonrotoclax 5 mg (1 tabl. at 5mg) Days 5-6 Sonrotoclax 10 mg (2 tabl. at 5mg) Days 7-8 Sonrotoclax 20 mg (1 tabl. at 20mg) Days 9-10 Sonrotoclax 40 mg (2 tabl. at 20mg) Days 11-12 Sonrotoclax 80 mg (1 tabl. at 80mg) Days 13-14 Sonrotoclax 160 mg (2 tabl. at 80mg) Days 15-16 Sonrotoclax 320 mg (4 tabl. at 80mg)
  Cycle 2-6: Day 1-21 Sonrotoclax 320 mg QD po
  Other Names: BGB-11417
  Arms: Tislelizumab + Zanubrutinib + Sonrotoclax

SUMMARY:
The aim of the CLL-RT1 trial is to evaluate the efficacy and safety of zanubrutinib (BGB-3111), a BTK inhibitor plus tislelizumab (BGB-A317), a PD1 inhibitor for treatment of patients with Richter Transformation

DETAILED DESCRIPTION:
Richter Transformation (RT) remains one of the biggest challenges in the treatment and management of CLL. While considerable progress has been made in the treatment of CLL, the prognosis of CLL patients with malignant disease transformation still is very poor and reported median OS is between 6 to 8 months. Conventional approaches with chemo- and chemoimmunotherapy have largely failed to improve response rates in RT patients. However, as the established treatment approach for de-novo Diffuse Large B Cell Lymphoma (DLBCL) is chemoimmunotherapy with a combination of Rituximab, Cyclophosphamid, Hydroxydaunorubicin, Vincristin and Prednisolon (R-CHOP), this has become the most commonly used regimen for lack of alternative strategies, despite poor efficacy. Patients being fit enough for allogeneic transplantation are undergoing this procedure after induction with R-CHOP. However, the majority of patients are not suitable for transplantation and relapse quickly. Hence, there is urgent need to improve therapy of RT by testing new compounds and combinations for treatment of this disease. Based on the available preclinical and preliminary clinical data on checkpoint inhibition plus Bruton's tyrosine (BTK) inhibition, the current trial will systematically assess the safety and toxicity of tislelizumab, a programmed cell death protein 1 (PD-1) inhibitor, plus zanubrutinib, a BTK inhibitor in patients with RT.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of CLL according to iwCLL criteria (Hallek et al, 2018)
2. Confirmed histopathological diagnosis of RT (diffuse large B-cell lymphoma or Hodgkin's lymphoma [Hodgkin's lymphoma only when not eligible for more in-tensive treatment])
3. Previously untreated RT or patients with objective response or non-tolerance to first-line RT treatment
4. Adequate bone marrow function as defined by:

   * Absolute neutrophil count (ANC) ≥ 1000/mm3, except for patients with bone marrow involvement in which ANC must be ≥ 500/mm3
   * Platelet ≥ 75,000/mm3, except for patients with bone marrow involvement in which the platelet count must be ≥ 30,000/mm3
5. Creatinine clearance ≥30ml/min calculated according to the modified formula of Cockcroft and Gault or directly measured with 24hr urine collection or an equivalent method.
6. Adequate liver function as indicated by a total bilirubin≤ 2 x, AST/ALT ≤ 2.5 x the institutional ULN value, unless directly attributable to the patient's CLL/RT or to Gilbert's Syndrome, in which case a max. total bilirubin ≤ 3 x and AST/ALT ≤ 5 x the institutional ULN value are required.
7. Negative serological testing for hepatitis B (HBsAg negative and anti-HBc nega-tive; patients positive for anti-HBc may be included if PCR for HBV DNA is negative and HBV-DNA PCR is performed every two months until 2 months af-ter last dose of zanubrutinib), negative testing for hepatitis-C RNA and negative HIV test within 6 weeks prior to registration
8. Age at least 18 years
9. ECOG performance status 0-2, ECOG 3 is only permitted if related to CLL or RT (e.g. due to anaemia or severe constitutional symptoms)
10. Life expectancy ≥ 3 months
11. Ability and willingness to provide written informed consent and to adhere to the study visit schedule and other protocol requirements

Exclusion Criteria:

1. Patients who did not respond to previous line of RT therapy (i.e. primary progressive patients)
2. Patients with more than one prior line of RT therapy
3. Allogenic stem cell transplantation within the last 100 days or signs of active GVHD after prior allogeneic stem cell transplantation within any time
4. Patients with confirmed PML
5. Uncontrolled autoimmune condition
6. Malignancies other than CLL currently requiring systemic therapies (unless the malignant disease is in a stable remission at the discretion of the treating phy-sician)
7. Uncontrolled infection currently requiring systemic treatment
8. Any comorbidity or organ system impairment rated with a CIRS (cumulative ill-ness rating scale) score of 4, excluding the eyes/ears/nose/throat/larynx organ system , or any other life-threatening illness, medical condition or organ system dysfunction that - in the investigator´s opinion could comprise the patients safety or interfere with the absorption or metabolism of the study drugs
9. Requirement of therapy with strong CYP3A4 inhibitors/ inducers
10. Requirement of therapy with phenprocoumon or other vitamin K antagonists.
11. Known active infection with HIV, or serologic status reflecting active hepatitis B or C infection as follows:

    * Presence of hepatitis B surface antigen (HBsAg) or hepatitis B core anti-body (HBcAb). Patients with presence of HBcAb, but absence of HBsAg, are eligible if hepatitis B virus (HBV) DNA is undetectable (< 20 IU), and if they are willing to undergo monitoring every 4 weeks for HBV reactivation.
    * Presence of hepatitis C virus (HCV) antibody. Patients with presence of HCV antibody are eligible if HCV RNA is undetectable.
12. Major surgery within 4 weeks of the first dose of study drug.
13. Any uncontrolled or clinically significant cardiovascular disease including the following:

    * Myocardial infarction within 6 months before screening
    * Unstable angina within 3 months before screening
    * New York Heart Association class III or IV congestive heart failure
    * History of clinically significant arrhythmias (eg, sustained ventricular tachy-cardia, ventricular fibrillation, torsades de pointes)
14. History of severe bleeding disorder such as hemophilia A, hemophilia B, von Willebrand disease, or history of spontaneous bleeding requiring blood trans-fusion or other medical intervention
15. History of stroke or intracranial hemorrhage within 6 months before first dose of study drug
16. Severe or debilitating pulmonary disease
17. Unable to swallow capsules or disease significantly affecting gastrointestinal function such as malabsorption syndrome, resection of the stomach or small bowel, bariatric surgery procedures, symptomatic inflammatory bowel disease, or partial or complete bowel obstruction
18. Use of investigational agents, e.g. monoclonal antibodies or other experimental drugs within clinical trials, which might interfere with the study drug within 28 days (or 5 times half-life [t1/2] of the compound, whichever is longer) prior to registration
19. Known hypersensitivity to tislelizumab, zanubrutinib, sonrotoclax or any of the excipients
20. Pregnant women and nursing mothers (a negative pregnancy test is required for all women of childbearing potential within 7 days before start of treatment)
21. Fertile men or women of childbearing potential unless:

    * surgically sterile or ≥ 2 years after the onset of menopause, or
    * willing to use two methods of reliable contraception including one highly ef-fective contraceptive method (Pearl Index <1) and one additional effective (barrier) method during study treatment and for 6 months after the end of study treatment.
22. Vaccination with a live vaccine <28 days prior to randomization
23. Legal incapacity
24. Prisoners or subjects who are institutionalized by regulatory or court order
25. Persons who are in dependence to the sponsor or an investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Estimated)
Dates: Start 2020-02-19 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) after induction therapy according to the refined Lugano Classification (Cheson et al, 2016) | 18 weeks
  Proportion of patients having achieved complete response (CR) or partial response (PR)

SECONDARY OUTCOMES:
ORR after induction therapy according to the IWCLL criteria (Hallek et al, 2018) | 18 weeks
  Proportion of patients having achieved complete response (CR) or partial response (PR)
ORR after consolidation therapy | 36 weeks
  Proportion of patients having achieved complete response (CR) or partial response (PR)
Progression-free Survival (PFS) | Up to 15 months
  Time from the date of registration to the date of first occurrence of disease progression or relapse (determined according to the IWCLL guidelines and Lugano classification) or death from any cause, whichever occurs first
Overall Survival (OS) | Up to 15 months
  Time from the date of registration to the date of death due to any cause
Time to Next Treatment (TTNT) | Up to 15 months
  Time from date of registration to the date of first subsequent CLL/RT treatment
Duration of response | Up to 15 months
  Time from the date of first documented response to the first occurrence of progression, relapse or death by any cause, whichever occurs first.
  Duration of response will be evaluated both according to the refined Lugano Classification as well as according to the IWCLL criteria. In the first case it will be calculated for patients with CR or PR, in the second case for patients with (clin.) CR, (clin.) CRi, PR, or PR-L.
Type, frequency, severity of adverse events (AEs) | Up to 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Eichhorst, Prof., Principal Investigator — Department I of Internal Medicine, University Hospital Cologne
Locations (11):
- Allgemeines Krankenhaus der Stadt Wien, Vienna, Austria
- Rigshospitalet, Copenhagen, Denmark
- Germany (9):
  - Charité Berlin, Berlin, State of Berlin
  - Uniklinik Köln, Cologne
  - Universitätsklinikum Carl Gustav Carus, Dresden
  - Universitätsklinikum Essen, Essen
  - Universitätsklinikum Schleswig-Holstein Campus Kiel, Kiel
  - H.O.T Praxis Landshut, Landshut
  - Brüderkrankenhaus St. Josef Paderborn, Paderborn
  - Universitätsmedizin Rostock, Rostock
  - Universitätsklinik Ulm, Ulm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Al-Sawaf O, Ligtvoet R, Robrecht S, Stumpf J, Fink AM, Tausch E, Schneider C, Boettcher S, Mikusko M, Ritgen M, Schetelig J, von Tresckow J, Vehling-Kaiser U, Gaska T, Wendtner CM, Chapuy B, Fischer K, Kreuzer KA, Stilgenbauer S, Staber P, Niemann C, Hallek M, Eichhorst B. Tislelizumab plus zanubrutinib for Richter transformation: the phase 2 RT1 trial. Nat Med. 2024 Jan;30(1):240-248. doi: 10.1038/s41591-023-02722-9. Epub 2023 Dec 9. PMID 38071379
- See also: Click here for more information about this study: CLL-RT1 (German CLL Study Group) — https://www.dcllsg.com/cll-rt1/